CLINICAL TRIAL: NCT03797729
Title: Early Initiation of Low Dose Tirofiban for Primary Percutaneous Coronary Intervention in Patients With ST-segment Elevation Myocardial Infarction.
Brief Title: Early Initiation of Low Dose Tirofiban for PPCI in STEMI Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRYIT
Record Dates: First submitted 2019-01-01; First posted 2019-01-09 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-01

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST Elevation Myocardial Infarction; Tirofiban; Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Tirofiban; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline
- Tirofiban (Experimental)
  Interventions: Drug: Tirofiban

INTERVENTIONS:
Drug: Tirofiban — Upon being diagnosed as ST Elevation Myocardial Infarction, if informed consent is obtained, patients start to receive Tirofiban(0.05mg/ml) intravenous drip in a dosage of 4ml/hour (patients weight<50kg) or 6ml/hour (patients weight > 50kg) lasting for 24 hours.
  Arms: Tirofiban
Drug: Normal saline — Upon being diagnosed as ST Elevation Myocardial Infarction, if informed consent is obtained, patients start to receive normal saline intravenous drip in a dosage of 4ml/hour (patients weight<50kg) or 6ml/hour (patients weight > 50kg) lasting for 24 hours.
  Other Names: Sodium Chloride Injection
  Arms: Normal saline

SUMMARY:
Anti-platelet therapy is a key point of acute myocardial infarction (AMI) treatment. Nowadays, dual anti-platelet therapy based on aspirin and ADP-P2Y12 receptor inhibitor is the preferred treatment before primary percutaneous coronary intervention (PPCI). Restricted by pharmacokinetic and pharmacodynamic characteristics, ADP-P2Y12 receptor inhibitors cannot take effect immediately after oral administration. However, platelet glycoprotein Ⅱb / Ⅲa inhibitors take effect faster. Previous clinical trials indicated that combination of full dose of glycoprotein Ⅱb / Ⅲa inhibitor and dual anti-platelet therapy reduced AMI related ischemia events but increased bleeding events significantly. The high dose of glycoprotein Ⅱb / Ⅲa inhibitor may be the key factor contributing to the increased bleeding events. Therefore, this study aims to evaluate the effectiveness and security of triple anti-platelet therapy based on a small dose of glycoprotein Ⅱb / Ⅲa inhibitor, aspirin and ADP-P2Y12 receptor inhibitor in AMI patients receiving PPCI.

ELIGIBILITY:
Inclusion Criteria:

* Time after onset of chest pain: ≥ 30 minutes and ≤ 24 hours;
* ST segment elevated ≥ 0.1mV in adjacent two or more leads;
* Scheduled for primary percutaneous coronary intervention without contraindications;
* Written informed consent is obtained.

Exclusion Criteria:

* Life expectancy ≤ 1 year;
* History of cerebral hemorrhage;
* History of stroke in 6 months;
* Active hemorrhage;
* Severe hepatic and renal dysfunction(ALT > 3 folds of upper limit of normal, eGFR < 30ml/min/1.73mm^2 or Scr > 200 mmol/L);
* Known hemorrhagic diseases;
* Known malignant tumour diseases；
* Active peptic ulcer disease;
* Blood platelet counts < 100×10^9/L;
* Blood hemoglobin < 90g/L;
* Pregnancy or lactation period；
* Take part in other intervention clinical trials；
* Investigators think not suitable to participate in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
TFG(TIMI flow grades) grade III: complete myocardial perfusion immediately after primary percutaneous coronary intervention detected by DSA(Digital Substraction Angiography). | Immediately after primary percutaneous coronary intervention.
  TIMI flow grades: grade III.
TMP(TIMI myocardial perfusion grades) grade III: complete myocardial perfusion immediately after primary percutaneous coronary intervention detected by DSA(Digital Substraction Angiography). | Immediately after primary percutaneous coronary intervention.
  TIMI myocardial perfusion grades: grade III.

SECONDARY OUTCOMES:
Remedial Tirofiban intravenous use during primary percutaneous coronary intervention procedure. | During the process of primary percutaneous coronary intervention.
  Remedial Tirofiban use during primary percutaneous coronary intervention.
ST segment | 90 minutes after primary percutaneous coronary intervention.
  The sum of the initial ST segment elevation drops 70% or more.
Myocardial microcirculation perfusion estimated by cardiac magnetic (CMR). | 7 days after primary percutaneous coronary intervention.
  Myocardial microcirculation perfusion estimated by cardiac magnetic resonance imaging.
Major adverse cardiovascular events(MACE), including a composite of all-cause death, nonfatal myocardial infarction, stroke, target vessel revascularization. | 30 days after primary percutaneous coronary intervention.
  Major adverse cardiovascular events, including a composite of all-cause death, nonfatal myocardial infarction, stroke, target vessel revascularization.

OTHER OUTCOMES:
Left ventricular ejection fraction (LVEF) assessed by transthoracic echocardiography. | 7 and 30 days after primary percutaneous coronary intervention.
  Left ventricular ejection fraction assessed by transthoracic echocardiography.
The serum microRNA expression pattern changes after primary percutaneous coronary intervention. | Pre-, 30 minutes, 3 hours and 24 hours after primary percutaneous coronary intervention.
  The microRNA expression pattern changes.
All the bleeding events assessed by bleeding academic research consortium(BARC) definition for bleeding) | 30 days after primary percutaneous coronary intervention.
  All the bleeding events assessed by bleeding academic research consortium(BARC) definition for bleeding)
Major bleeding events assessed by TIMI bleeding criteria. | 30 days after primary percutaneous coronary intervention.
  Any intracranial bleeding (excluding microhemorrhages <10 mm evident only on gradient-echo MRI); Clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥ 5 g/dL; Fatal bleeding (bleeding that directly results in death within 7 d).
Severe or life-threatening and moderate bleeding events assessed by GUSTO bleeding criteria. | 30 days after primary percutaneous coronary intervention.
  GUSTO bleeding criteria:Severe or life-threatening :
  Intracerebral hemorrhage ; Resulting in substantial hemodynamic compromise requiring treatment.
  Moderate:
  Requiring blood transfusion but not resulting in hemodynamic compromise.
  Mild :
  Bleeding that does not meet above criteria.
Major bleeding events assessed by international society on thrombosis and haemostasis(ISTH) bleeding criteria. | 30 days after primary percutaneous coronary intervention.
  Fatal bleeding and/or symptomatic bleeding in a critical area or organ such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing hemoglobin drop of 20 g/L or more, and/or blood transfusion of 2 units or more
Adverse events and severe adverse events. | 30 days after primary percutaneous coronary intervention.
  Adverse events and severe adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Juying Qian, MD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No